CLINICAL TRIAL: NCT06843330
Title: Are Portable Lactate Monitoring Devices Accurate in Patients With Glycogen Storage Disease Ia When Compared to Blood Serum Lactates?
Brief Title: Accuracy of Lactate Meter in GSDIa
Status: Recruiting | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Jewish Community Foundation (Unknown)
Responsible Party: Principal Investigator, Rebecca Riba-Wolman, Principal Investigator, Connecticut Children's Medical Center
Other Study IDs: 23-137
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Glycogen Storage Disease Type Ia
Keywords: Glycogen Storage Disease type Ia; Blood lactate; Glycogen Storage Disease Ia blood glucose; GSD I; GSDIa; Blood glucose; Accu chek glucometer; Lactate plus
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: blood glucose meter; blood lactate meter — Blood lactate level measured by finger-stick with over the counter meter. Blood glucose level measured by finger-stick.

SUMMARY:
The goal of this observational study is to determine if home lactate meters (both capillary and serum sample) are accurate, compared to lab serum lactate in a population of patients with glycogen storage disease type 1a and to determine if the Accu Chek Guide glucometer (capillary sample) is accurate, in a population of patients with glycogen storage disease type 1a.

DETAILED DESCRIPTION:
The goal of this observational study is to determine if home lactate meters (both capillary and serum sample) are accurate, within 20% of lab serum lactate reading 95% of the time, in a population of patients with glycogen storage disease type 1a and to determine if the Accu Chek Guide glucometer (capillary sample) is accurate, within 20% of lab serum glucose reading 95% of the time, in a population of patients with glycogen storage disease type 1a.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed/confirmed (by liver biopsy or genetic testing) Glycogen Storage Disease Type Ia (ICD 10 code: E74.01).
* Connecticut Children's Emergency Department visit and/or admission to Connecticut Children's during time study is active
* For pediatric participants: Ability of child's parent/legal guardian to understand and the willingness to sign a written informed consent document
* For adults: Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with Glycogen storage disease unspecified 74.00, or Ib
* Patients not meeting inclusion criteria

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients of Connecticut Children's birth to age 60 years with diagnosed Glycogen Storage Disease Type Ia, that are seen in clinic between 7/2020 - 7/2024, or that present to emergency room or are admitted to Connecticut Children's for surgery, acute illness or dose titration admission.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Home lactate meter accuracy in GSDIa compared with lab lactate | Every 1-3 hours for a maximum 33 hours
  Lactate level via point of care finger-stick and lab draw

SECONDARY OUTCOMES:
Glucometer accuracy in GSDIa compared with lab lactate | Every 1-3 hours for a maximum 33 hours
  Glucose level via finger-stick and lab draw

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No